CLINICAL TRIAL: NCT01431599
Title: Two Week-course Preoperative Chemoradiotherapy Followed by Delayed Operation for Rectal Cancer: Phase II Multicenter Clinical Trial (KROG 11-02)
Brief Title: Short-course Preoperative Chemoradiotherapy for Rectal Cancer
Acronym: KROG 11-02
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jong Hoon Lee (Other)
Collaborators: Seoul National University Hospital (Other); Samsung Medical Center (Other); National Cancer Center, Korea (Other Government)
Responsible Party: Sponsor-Investigator, Jong Hoon Lee, Dr., Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KROG 11-02
Record Dates: First submitted 2011-09-06; First posted 2011-09-09 (Estimated); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Rectal Cancer
Keywords: Locally advanced rectal cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- short-course (Experimental)
  Interventions: Radiation: short-course radiation

INTERVENTIONS:
Radiation: short-course radiation — 33Gy/10 fractions

SUMMARY:
The purpose of this study is to evaluate the early clinical outcome of the short-course preoperative chemoradiotherapy, 33Gy/10 fx and delayed operation after chemoradiation, the investigators initiated the clinical trial of KROG 11-02.

ELIGIBILITY:
Inclusion Criteria:

1. histologically confirmed adenocarcinoma
2. distal margin of the tumor located < 8 cm above the anal verge
3. cT3-4 or cN+ classification as determined by endorectal ultrasonography (EUS) and CT
4. patient older than age 18 years
5. Karnofsky performance score >= 70

Exclusion Criteria:

1. distant metastasis identified during staging workup
2. previous or concurrent malignancy
3. pregnant or breast-feeding women
4. impending rectal obstruction
5. familial adenomatous polyposis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-10 (Actual); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
downstaging effect of tumor | an expected average of 6 weeks after chemoradiation
  Comparison of clinical T staging and pathologic T staging example> cT4 --> pT1 after chemoradiation: down staging (+)

SECONDARY OUTCOMES:
bladder and small bowel toxicity after chemoradiation | Participants will be followed for an expected average of 3 months after chemoradiation
  The incidence of grade 3 or higher small bowel and bladder toxicity according to the RTOG and EORTC toxicity criteria (reference: Cox JD et al. Int J Radiat Oncol Biol Phys. 1995 Mar 30;31(5):1341-6)

CONTACTS AND LOCATIONS:
Overall Officials: Hong Seok Jang, MD, Principal Investigator — Department fo Radiation Oncology, Seoul St. Mary's Hospital
Locations (3):
- South Korea (3):
  - National Cancer Center, Korea, Goyang
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul

REFERENCES:
- [Background] Swedish Rectal Cancer Trial; Cedermark B, Dahlberg M, Glimelius B, Pahlman L, Rutqvist LE, Wilking N. Improved survival with preoperative radiotherapy in resectable rectal cancer. N Engl J Med. 1997 Apr 3;336(14):980-7. doi: 10.1056/NEJM199704033361402. PMID 9091798
- [Background] Gerard A, Buyse M, Nordlinger B, Loygue J, Pene F, Kempf P, Bosset JF, Gignoux M, Arnaud JP, Desaive C, et al. Preoperative radiotherapy as adjuvant treatment in rectal cancer. Final results of a randomized study of the European Organization for Research and Treatment of Cancer (EORTC). Ann Surg. 1988 Nov;208(5):606-14. doi: 10.1097/00000658-198811000-00011. PMID 3056288
- [Derived] Lee JH, Kim JG, Oh ST, Lee MA, Chun HG, Kim DY, Kim TH, Kim SY, Baek JY, Park JW, Oh JH, Park HC, Choi DH, Park YS, Kim HC, Chie EK, Jang HS. Two-week course of preoperative chemoradiotherapy followed by delayed surgery for rectal cancer: a phase II multi-institutional clinical trial (KROG 11-02). Radiother Oncol. 2014 Jan;110(1):150-4. doi: 10.1016/j.radonc.2013.11.013. Epub 2014 Jan 7. PMID 24411228